CLINICAL TRIAL: NCT06382090
Title: The Effect of Laughter Yoga on Premenstrual Syndrome in Adolescents
Brief Title: Premenstrual Syndrome and Laughter Yoga
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Burcu Bakırlıoğlu, Research Assistant, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PamukkaleU-SBE-BB-01
Record Dates: First submitted 2024-04-20; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Premenstrual Syndrome; Laughter
Keywords: Laughter Yoga; Premenstrual Syndrome; Adolescent
MeSH Terms: conditions — Premenstrual Syndrome; Laughter | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Two groups: comparative experiment and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter yoga (Experimental): Premenstrual syndrome scale will be applied to adolescents as a pre-test. 34 randomly selected students who pass the cutoff score on this scale will form the experimental group. A total of 10 sessions of laughter yoga will be performed for this group, twice a week for 5 weeks. At the end of the tenth session, the premenstrual syndrome scale will be re-applied to the experimental group as a post-test.
  Interventions: Other: Laughter yoga
- Control (No Intervention): Premenstrual syndrome scale will be applied to adolescents as a pre-test. 34 randomly selected students who pass the cutoff score on this scale will form the control group. No intervention will be applied to this group. At the end of five weeks, the premenstrual syndrome scale will be applied again to the control group as a post-test.

INTERVENTIONS:
Other: Laughter yoga — This practice, which includes deep breathing exercises and laughter exercises, takes approximately 45 minutes. The sessions will be conducted by the principal investigator.
  Arms: Laughter yoga

SUMMARY:
In addition to physical and emotional effects, premenstrual syndrome can negatively affect the participation in classes, school success, social activities and family relationships of young adolescents in high school. Many non-pharmacological treatments have been found to improve premenstrual syndromes in adolescents. Laughter yoga, one of these methods, is a practice consisting of deep breathing exercises and laughter exercises. Laughter yoga has been studied in different sample groups (elderly people, nurses, dialysis patients, etc.) and positive results have been obtained. In this study, the effect of laughter yoga on premenstrual symptoms in adolescents will be examined.

DETAILED DESCRIPTION:
According to the Nursing Interventions Classification (NIC), laughter therapy, one of the interventions used in nursing care, appears as a universal approach. Laughter therapy is defined as facilitating the patient's perception, appreciation, and expression of what is funny, entertaining, or ridiculous in order to build relationships, reduce tension, release anger, facilitate learning, or cope with painful emotions. Laughter therapy, which is applied without using humor, generally includes exercises such as clapping, dancing, and vocalizing laughter-like sounds such as "hoho-hahaha", but it can also include non-laughter elements such as breathing and relaxation exercises. Laughter Yoga is a specific example of non-humorous laughter therapy; It includes yoga exercises such as laughing exercises, clapping, breathing and relaxation exercises. In studies conducted in the pediatric population, laughter yoga has been shown to improve stress, pain, self-esteem , anxiety, hopelessness. Has been found to provide positive improvements in depression and psychological resilience.

The menstrual cycle, which is one of the most important signs of the functioning of the reproductive system, is associated with signs and symptoms that cause physical and psychological problems. Premenstrual Syndrome (PMS) refers to a set of recurrent symptoms that begin at the end of the luteal phase of the menstrual cycle (5-7 days before menstruation) and end in the follicular phase (2-4 days after menstruation). Many women cannot cope with symptoms such as emotional changes, irritability, lack of concentration, depressive mood or insomnia that occur during this period. For this reason, premenstrual symptoms can negatively affect adolescents' participation in classes, school success, social activities and family relationships. In addition to pharmacological agents, non-pharmacological methods such as reflexology, acupuncture, acupressure, cognitive-behavioral approaches and massage therapy have been used in recent years to cope with premenstrual syndrome.

PMS is an important health problem that includes complex symptoms and negatively affects women's quality of life. In order to cope with these symptoms, PMS needs to be addressed multidimensionally. This study aimed to investigate the effect of laughter therapy in coping with premenstrual syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research
* Having a regular menstrual cycle (menstruation every 21-35 days and without complaints of intermittent bleeding) for the last 6 months
* Not receiving medical treatment for PMS

Exclusion Criteria:

* Not agreeing to participate in the research
* Having had any surgical operation in the last 3 months
* Presence of a chronic disease (asthma, DM, etc.)
* Presence of gynecological disease
* Using hormonal contraception (such as oral contraceptives and injections).

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2024-04-26 (Estimated); Primary Completion 2024-05-24 (Estimated); Study Completion 2025-05-24 (Estimated)

PRIMARY OUTCOMES:
Premenstrual Symptom Scale | 5 weeks
  Premenstrual Syndrome Scale is a five-point Likert type scale with 44 items. In the application of PMSS, as stated in the instruction at the beginning, after reading the item, marking is made according to whether this situation is "one week before menstruation", taking into account the degrees to the right of the relevant item. In scoring the scale, the "Never" option is evaluated as 1 point, the "Very little" option is evaluated as 2 points, the "Sometimes" option is evaluated as 3 points, the "Often" option is evaluated as 4 points and the "Always" option is evaluated as 5 points. The scale has a total of nine subscales: Depressive Affect, Anxiety, Fatigue, Irritability, Depressive Thoughts, Pain, Appetite Changes, Sleep Changes and Bloating. The higher the score, the more intense the premenstrual syndrome symptoms are considered.

IPD SHARING:
Plan to Share IPD: No